CLINICAL TRIAL: NCT06712342
Title: Effects of Upper Extremity-Focused Neuromuscular Exercise Training on Physical and Cognitive Functions in People With Multiple Sclerosis (NExTUp)
Brief Title: Effects of Upper Extremity-Focused Neuromuscular Training in People With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Uğur OVACIK, PT, MSc, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/125
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; exercise; function; upper extremity; neuromuscular exercise training; manual dexterity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEG (Experimental): Upper Extremity Focused Neuromuscular Exercise Training
  Interventions: Other: Neuromuscular Exercise Training
- CEG (Active Comparator): Traditional Upper Extremity Exercise Training
  Interventions: Other: Conventional Exercise Training
- CG (No Intervention): Control Group

INTERVENTIONS:
Other: Neuromuscular Exercise Training — This group will receive neuromuscular exercise training with 60-75 minute sessions per day, 2 days a week, for 8 weeks.
  Warm-up Program - 5 minutes Postural Control-Weight Transfer - 10-15 minutes Strength Training - 30-35 minutes Proprioception - Coordination - Reaction Speed 10-15 minutes Cool-down Program - 5 minutes
  Arms: NEG
Other: Conventional Exercise Training — This group will be given traditional strength exercise training consisting of 60-75 minute sessions per day, 2 days per week for 8 weeks.
  Warm-up Program - 5 minutes Strength Training - 30-35 minutes Manuel Dexterity - 15-20 minutes Cool-down Program - 5 minutes
  Arms: CEG

SUMMARY:
The effectiveness of upper extremity focused neuromuscular exercise training in early stage people with MS will be investigated. People with MS enrolled in the study will be randomly assigned to three groups: Neuromuscular Exercise Group (NEG), Conventional Exercise Group (CEG), and Control Group (CG). All three groups will be assessed with primary and secondary outcome measures at baseline, week 8, and week 12. NEG, CEG, and CG will be initially assessed for upper extremity function, cognitive function, lower extremity function, grip strength, proximal muscle strength, sensation, coordination, fatigue, postural sway, and core muscle strength and endurance. Then, NEG will receive clinically supervised upper extremity focused neuromuscular exercise training with a minimum of 60 minutes of session time, 2 days a week for 8 weeks. This exercise training includes steps for postural control, weight transfer, proximal and distal muscle strengthening, proprioception, coordination and reaction speed. Similarly, CEG will receive clinically supervised traditional upper extremity exercise training, twice a week for 8 weeks, with a minimum of 60 minutes of session time. This exercise training includes strengthening with the band and manuel dexterity exercises. In both groups, stretching and mobility exercises will be added to the warm-up and cool-down exercises before and after the program. During this process, CG will be on the waiting list. At the end of 8 weeks, all three groups will be re-evaluated. After the exercise training, follow-up will be done and evaluations will be repeated in the 12th week. This study will provide evidence on the effects of upper extremity-focused neuromuscular exercise training on physical and cognitive functions in early-stage people with MS compared to traditional treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS according to McDonald criteria,
* 18-64 years
* RRMS,
* EDSS < 4,
* Minimal or moderate upper extremity involvement

Exclusion Criteria:

* Having an attack in the last three months,
* Mini Mental Test <24 or visual deficit,
* Other medical conditions accompanying MS (cardiac, orthopedic or rheumatic, etc.),
* Being pregnant or breastfeeding,
* Doing regular exercise - receiving physiotherapy,
* Having spasticity of 2 or more in the upper extremity

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test | At the beginning, at the end of 8 weeks and 12 weeks
  To assess unilateral function of the upper extremity
Minnesota Manual Dexterity Test | At the beginning, at the end of 8 weeks and 12 weeks
  To assess bilateral upper extremity function
Manual Ability Measure-36 | At the beginning, at the end of 8 weeks and 12 weeks
  To assess upper extremity function. A higher score indicates better hand function.
Timed 25-Foot Walk | At the beginning, at the end of 8 weeks and 12 weeks
  To assess lower extremity function
Symbol Digit Modalities Test | At the beginning, at the end of 8 weeks and 12 weeks
  To assess cognitive function
Hand Dynamometer | At the beginning, at the end of 8 weeks and 12 weeks
  To assess hand grip strength

SECONDARY OUTCOMES:
Hand Held Dynamometer | At the beginning, at the end of 8 weeks and 12 weeks
  To assess elbow muscle strength
Biodex Balance System | At the beginning, at the end of 8 weeks and 12 weeks
  To assess postural sway
Laser-pointer Assisted Angle Reproduction Test | At the beginning, at the end of 8 weeks and 12 weeks
  To assess of shoulder proprioception
Finger Tapping Test | At the beginning, at the end of 8 weeks and 12 weeks
  To assess upper extremity coordination
Fatigue Severity Scale | At the beginning, at the end of 8 weeks and 12 weeks
  To assess fatigue severity. A high score indicates high fatigue severity.
Plank | At the beginning, at the end of 8 weeks and 12 weeks
  To assess core muscle endurance
Curl-up | At the beginning, at the end of 8 weeks and 12 weeks
  To assess core muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Ovacık, Principal Investigator — Istanbul Aydın University; Ela Tarakcı, Study Director — Istanbul University - Cerrahpasa